CLINICAL TRIAL: NCT01510327
Title: PLATINUM: A Prospective, Randomized, Multicenter Trial to Assess an Everolimus-Eluting Coronary Stent System (PROMUS Element™) for the Treatment of up to Two De Novo Coronary Artery Lesions - Pharmacokinetics Sub-trial
Brief Title: PLATINUM Trial to Assess the PROMUS Element Stent System for Treatment of De Novo Coronary Artery Lesions-Pharmacokinetics (PLATINUM PK)
Acronym: PLATINUM PK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2046B
Record Dates: First submitted 2011-12-21; First posted 2012-01-16 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stents; DES; atherosclerotic
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; thienopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PROMUS Element (Experimental): Patients who received the PROMUS Element everolimus-eluting stent (EES) implanted using standard percutaneous coronary intervention (PCI) technique. Total loaded dose of everolimus per stent is dependent on stent size and in this study the administered dose ranged from 60.1 µg to 138.6 µg per stent. Note that the total dose of everolimus administered to a patient is based on the number of stents received and the size of the stent(s). The total dose received per patient ranged from 60.1 µg to 197.8 µg.
  Interventions: Device: PROMUS Element Everolimus-Eluting Coronary Stent System; Drug: Aspirin; Drug: Thienopyridine

INTERVENTIONS:
Device: PROMUS Element Everolimus-Eluting Coronary Stent System — PROMUS Element is a device/drug combination product composed of two components, a device (coronary stent system including a platinum chromium stent platform) and a drug product (a formulation of everolimus contained in a polymer coating).
Drug: Aspirin — Patients are required to take aspirin indefinitely after stent implant. It is recommended that aspirin 162-325 mg daily be given for at least 6 months after stent placement and that aspirin 75-162 mg daily be given indefinitely thereafter.
Drug: Thienopyridine — Patients must be treated with one of the following thienopyridines for at least 6 months following the index procedure: clopidogrel 75 mg daily; or ticlopidine 250 mg twice daily; or prasugrel (outside the United States and if approved at the time of the procedure). If used, the prescribed dose should be in accordance with approved country-specific labeling. In patients not at high risk of bleeding, thienopyridine treatment should continue for at least 12 months after stent implant.
  Other Names: A brand name for clopidogrel is PLAVIX.; A brand name for ticlopidine is TICLID.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the PROMUS Element™ Everolimus-Eluting Coronary Stent System for the treatment of patients with up to 2 de novo atherosclerotic coronary artery lesions. The lesions are located in vessels that are average-sized.

DETAILED DESCRIPTION:
The wide-spread use of drug-eluting stents (DES) has evolved as standard of care in de novo lesions. The proposed study will evaluate the safety and effectiveness of PROMUS Element for the treatment of de novo atherosclerotic lesions in native coronary arteries. The study design is consistent with the draft guidance for industry titled, "Coronary Drug-Eluting Stents - Nonclinical and Clinical Studies" (March 2008).

During the trial, thienopyridines must be administered according to the 2007 American College of Cardiology (ACC)/American Heart Association (AHA)/Society for Cardiovascular Angiography and Interventions (SCAI) guidelines, which recommended that clopidogrel (75 mg daily) or ticlopidine (250 mg twice daily) be prescribed after stent implantation for at least 6 months in all patients, and for at least 12 months in patients who are not at high risk of bleeding. For sites in the United States, the use of prasugrel is not allowed as part of the PLATINUM Clinical Trial. For sites in other countries, prasugrel may be prescribed according to its approved dosing in countries in which it is available. For patients taking aspirin daily a loading dose is recommended; for patients who have not been taking aspirin daily, aspirin must be administered as a loading dose. Patients continue to take aspirin indefinitely to reduce the risk of thrombosis.

This PLATINUM Pharmacokinetics (PK) study is a sub-trial associated with the PLATINUM Workhorse Randomized Controlled Trial, which is registered under NCT00823212. PLATINUM PK was designed to evaluate the elution of everolimus from the PROMUS Element everolimus-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient (or legal guardian) understands study requirements and treatment procedures and provides written informed consent before any study-specific tests or procedures are performed
* For patients less than 20 years of age enrolled at a Japanese site, patient and patient's legal representative must provide written informed consent before any study-specific tests or procedures are performed
* Patient is eligible for percutaneous coronary intervention (PCI)
* Patient has documented stable angina pectoris or documented silent ischemia; or unstable angina pectoris
* Patient is an acceptable candidate for coronary artery bypass grafting (CABG)
* Patient has a left ventricular ejection fraction (LVEF) >=30% as measured within 30 days prior to enrollment
* Patient is willing to comply with all protocol-required follow-up evaluations

Angiographic Inclusion Criteria (visual estimate):

• Target lesion must be a de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter (RVD) >=2.50 mm and <=4.25 mm. Target lesion length must measure (by visual estimate) <=24 mm. Target lesion must be in a major coronary artery or branch with visually estimated stenosis >=50% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow >1.

Exclusion Criteria:

* Patient has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute myocardial infarction (MI)
* Patient has had a known diagnosis of recent MI (ie, within 72 hours prior to index procedure) and has elevated enzymes at time of index procedure as follows.

  * Patients are excluded if any of the following criteria are met at time of the index procedure.

    * If creatine kinase-myoglobin band(CK-MB) >2× upper limit of normal (ULN), the patient is excluded regardless of CK Total.
    * If CK-MB is 1-2× ULN, the patient is excluded if the CK Total is >2× ULN.
  * If CK Total/CK MB are not used and Troponin is, patients are excluded if the following criterion is met at time of index procedure.

    * Troponin >1× ULN with at least one of the following.
    * Patient has ischemic symptoms and ECG changes indicative of ongoing ischemia (eg, >1 mm ST segment elevation or depression in consecutive leads or new left bundle branch block [LBBB]);
    * Development of pathological Q waves in the ECG; or
    * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

Note: For patients with unstable angina or patients who have had a recent MI, CK Total/CK MB (or Troponin if CK Total/CK MB are not used) must be documented prior to enrolling/randomizing the patient.

* Patient has received an organ transplant or is on a waiting list for an organ transplant
* Patient is receiving or scheduled to receive chemotherapy within 30 days before or after index procedure
* Patient is receiving oral or intravenous immunosuppressive therapy (ie, inhaled steroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (eg, human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
* Patient is receiving chronic (>=72 hours) anticoagulation therapy (eg, heparin, coumadin) for indications other than acute coronary syndrome
* Patient has platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Patient has white blood cell (WBC) count <3,000 cells/mm3
* Patient has documented or suspected liver disease, including laboratory evidence of hepatitis
* Patient is on dialysis or has known renal insufficiency (ie, estimated creatinine clearance <50 ml/min by the Cockcroft Gault formula, or [(140-age)*lean body weight (in kg)]/[plasma creatinine (mg/dl)*72])
* Patient has history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Target vessel(s) or side branch has been treated with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to index procedure
* Target vessel(s) has been treated within 10 mm proximal or distal to target lesion (by visual estimate) with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) at any time prior to index procedure
* Non-target vessel or side branch has been treated with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 24 hours prior to index procedure
* Planned or actual target vessel(s) treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter immediately prior to stent placement
* Planned PCI or CABG after index procedure
* Patient previously treated at any time with coronary intravascular brachytherapy
* Patient has a known allergy to the study stent system or protocol-required concomitant medications (eg, stainless steel, platinum, cobalt, chromium, nickel, tungsten, acrylic, fluoropolymers, everolimus, thienopyridines, aspirin, contrast) that cannot be adequately premedicated
* Patient has active peptic ulcer or active gastrointestinal (GI) bleeding
* Patient has one of the following.

  * Other serious medical illness (eg, cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
  * Current problems with substance abuse (eg, alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with protocol or confound data interpretation
* Patient is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Patient intends to participate in another investigational drug or device clinical trial within 12 months after index procedure
* Patient with known intention to procreate within 12 months after index procedure (Women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure.)
* Patient is a woman who is pregnant or nursing (A pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
* Patient has more than 2 target lesions, or more than 1 target lesion and 1 non-target lesion, which will be treated during the index procedure

Angiographic Exclusion Criteria (visual estimate):

* Target lesion meets any of the following criteria:

  * Aorto-ostial location (ie, lesion located within 5 mm of ostium by visual estimate)
  * Left main location
  * Located within 5 mm of origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery by visual estimate
  * Located within a saphenous vein graft or arterial graft
  * Will be accessed via a saphenous vein graft or arterial graft
  * Involves a side branch >=2.0 mm in diameter by visual estimate
  * Involves a clinically significant side branch <2.0 mm in diameter by visual estimate that has a clinically significant stenosis at the ostium
  * TIMI flow 0 (total occlusion) or TIMI flow 1 prior to wire crossing
  * Excessive tortuosity proximal to or within the lesion
  * Extreme angulation proximal to or within the lesion
  * Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified by visual estimate
  * Restenotic from previous intervention
  * Thrombus, or possible thrombus, present in target vessel
* Non-target lesion to be treated during the index procedure meets any of the following criteria:

  * Located within the target vessel
  * Located within a bypass graft (venous or arterial)
  * Left main location
  * Chronic total occlusion
  * Involves a complex bifurcation (eg, bifurcations requiring treatment with more than 1 stent)
  * Restenotic from previous intervention
* Patient has unprotected left main coronary artery disease (>50% diameter stenosis)
* Patient has protected left main coronary artery disease and a target lesion in the LAD or LCX
* Patient has an additional clinically significant lesion(s) in target vessel for which an intervention within 12 months after the index procedure is likely to be required
* Patient has 2 target lesions in the same vessel that are separated by less than 15 mm (by visual estimate) Note: Multiple focal stenoses will be considered as a single lesion if they can be completely covered with 1 stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M. Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (5):
- United States (2):
  - Medical Center of the Rockies (Loveland), Loveland, Colorado
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
- Japan (3):
  - Saiseikai Yokohama-City Eastern Hospital, Yokohama, Kanagawa
  - Sakakibara Heart Institute, Japan Research Promotion Society for Cardiovascular Diseases, Fuchu-shi, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo-to

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 9, 2009 to February 9, 2010 there were 11 patients enrolled at 2 investigative sites in the United States and 11 patients enrolled at 3 sites in Japan. All enrolled patients received a PROMUS Element study stent.
Groups:
- PROMUS Element: Patients who received the PROMUS Element everolimus-eluting stent (EES) implanted using standard percutaneous coronary intervention (PCI) technique
Period: Overall Study
Arm/Group | PROMUS Element
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 11
  Japan | 11
Cardiac History [Number; unit: Participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participants
    Previous Percutaneous Coronary Intervention (PCI) | 9
    Previous Coronary Artery Bypass Graft (CABG) | 2
    Previous Myocardial Infarction (MI) | 4
    Stable Angina | 15
    Unstable Angina | 2
    Silent Ischemia | 5
    History of Multivessel Disease | 9
Cardiac History - Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Percent (of blood emptied)] — Left ventricular ejection fraction (LVEF) is an assessment (fraction) of the amount of blood emptied from the left ventricle during systolic contraction, which is indicative of global ventricular function.
  Percent (of blood emptied) | 59.64 (10.09)
Height [Mean (Standard Deviation); unit: Centimeters] | 165.57 (12.55)
Weight [Mean (Standard Deviation); unit: Kilograms] | 73.68 (19.60)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.52 (4.79)
Cardiac Risk Factors [Number; unit: Participants] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participants
    Smoking, ever | 14
    Medically Treated Diabetes | 5
    Hyperlipidemia Requiring Medication | 16
    Hypertension Requiring Medication | 18
Comorbidities [Number; unit: Participants] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participants
    History of Transient Ischemic Attack | 2
    History of Cerebrovascular Accident | 3
    History of Peripheral Vascular Disease | 2
    History of Renal Disease | 0
Lesion Characteristic: Target Lesion Vessel [Number; unit: Lesions] — 24 lesions in 22 participants were treated.
  Lesions
    Left Anterior Descending Artery | 4
    Left Circumflex Artery | 7
    Right Coronary Artery | 13
Lesion Characteristic: Lesion Location [Number; unit: Participants] — 24 lesions treated in 22 participants.
  Participants
    Proximal | 9
    Mid | 13
    Distal | 2
Lesion Characteristics: Reference Vessel Diameter, Minimum Lumen Diameter, Length [Mean (Standard Deviation); unit: millimeters] — There were 24 lesions treated in 22 participants.
  millimeters
    Reference Vessel Diameter | 2.64 (0.46)
    Minimum Lumen Diameter | 0.73 (0.38)
    Lesion Length | 12.11 (4.69)
Lesion Characteristic-Percent Diameter Stenosis [Mean (Standard Deviation); unit: Percent] — There were 24 lesions treated in 22 participants.
  Percent | 73.15 (11.24)
Lesion Characteristics [Number; unit: Lesions] — There were 24 lesions treated in 22 participants. The same lesion may be included in more than one category, therefore the number of lesions for this baseline measure does not equal the total number of lesions in the group.
  Lesions
    Eccentric Lesion | 13
    Bend >45 Degrees | 13
    Bend >90 Degrees | 2
    Tortuosity, any | 1
    Calcification, any | 4
    Bifurcation | 1
Lesion Characteristics: American College of Cardiology (ACC)/American Heart Association (AHA) Class [Number; unit: Lesions] — Type A: minimally complex, readily accessible, non angulated, smooth contour, little to no calcification, less than totally occlusive, not ostial in location, no major side branch involvement, absence of thrombus.
  Type B: moderately complex, eccentric, moderate tortuosity and angulation, moderate or heavy calcification, total occlusion < 3 months old, ostial in location, presence of thrombus; type B1 has one adverse characteristic and B2 has ≥2. Type C: severely complex, diffuse, excessive tortuosity and angulation, total occlusions > 3 months old, degenerated vein grafts and friable lesions.
  Lesions
    A | 1
    B1 | 4
    B2 | 15
    C | 4
Lesion Characteristic - Pre-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: Lesions] — 24 lesions treated in 22 participants. Thrombolysis In Myocardial Infarction (TIMI)0 - No perfusion; TIMI 1 - Penetration with minimal perfusion; TIMI 2 - Partial perfusion; TIMI 3 - Complete perfusion
  Lesions
    TIMI 0 | 0
    TIMI 1 | 0
    TIMI 2 | 0
    TIMI 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Everolimus Blood Concentration (Cmax)
Description: Venous blood draw up to 24 hours prior to implantation of the first study stent (predose time point) and at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours after completion of implantation of the last study stent
Time Frame: Predose <24 hours; post dose at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours
Population: The analysis groups reported here had 3 or more subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Everolimus Dose of 95.4 µg; Everolimus Dose of 102.4 µg; Everolimus Dose of 138.6 µg: Patients who received the PROMUS Element everolimus-eluting stent (EES) implanted using standard percutaneous coronary intervention (PCI) technique; total dose of everolimus administered is based on the number of stents received and the size of the stents
Arm/Group | Everolimus Dose of 95.4 µg | Everolimus Dose of 102.4 µg | Everolimus Dose of 138.6 µg
Number analyzed (Participants) | 4 | 7 | 3
ng/mL | 0.71 (0.09) | 0.67 (0.15) | 0.91 (0.20)

2. Secondary Outcome: Area Under the Concentration Versus Time Curve (AUC 0-t) Everolimus
Description: Venous blood draw up to 24 hours prior to implantation of the first study stent (predose time point) and at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours after completion of implantation of the last study stent; t is the last time at which concentration can be quantified
Time Frame: Predose <24 hours; post dose at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours
Population: The analysis groups reported here had 3 or more subjects.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Everolimus Dose of 95.4 µg; Everolimus Dose of 102.4 µg; Everolimus Dose of 138.6 µg: Patients who received the PROMUS Element everolimus-eluting stent (EES) implanted using standard percutaneous coronary intervention (PCI) technique; the dose of everolimus is based on the number and sizes of stents implanted
Arm/Group | Everolimus Dose of 95.4 µg | Everolimus Dose of 102.4 µg | Everolimus Dose of 138.6 µg
Number analyzed (Participants) | 4 | 7 | 3
ng*hr/mL | 7.27 (4.97) | 6.45 (5.26) | 10.87 (7.36)

3. Secondary Outcome: Area Under the Concentration Versus Time Curve (AUC 0-24), Everolimus
Description: as for outcome 1
Time Frame: Predose <24 hours; post dose at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours
Population: The analysis groups reported here had 3 or more subjects.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Everolimus Dose of 95.4 µg | Everolimus Dose of 102.4 µg | Everolimus Dose of 138.6 µg
Number analyzed (Participants) | 4 | 7 | 3
ng*hr/mL | 6.83 (2.03) | 6.14 (1.10) | 9.51 (0.64)

4. Secondary Outcome: Area Under the Concentration Versus Time Curve (AUC 0-infinity) Everolimus
Description: Venous blood draw up to 24 hours prior to implantation of the first study stent (predose time point), 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours after implantation of the last study stent.
Time Frame: Predose <24 hours; post dose at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours
Population: Analysis groups have ≥3 subjects. Everolimus concentrations declined rapidly in all subjects; AUC0-∞ could be inaccurately determined for a subset of samples. AUC0-∞ determined by extrapolation of terminal phase. Concentrations not above detection limit in the terminal phase for enough time points for most subjects to accurately determine AUC0-∞.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Everolimus Dose of 95.4 µg | Everolimus Dose of 102.4 µg | Everolimus Dose of 138.6 µg
Number analyzed (Participants) | 4 | 7 | 3
ng*hr/mL | 19.26 (11.69) | 12.95 (2.05) | 60.74 (25.95)

5. Secondary Outcome: Time of Occurrence of Maximum Everolimus Concentration (Tmax)
Description: as for outcome 1
Time Frame: Predose <24 hours; post dose at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours
Population: Analysis groups reported here had 3 or more subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Everolimus Dose of 95.4 µg | Everolimus Dose of 102.4 µg | Everolimus Dose of 138.6 µg
Number analyzed (Participants) | 4 | 7 | 3
hours | 0.47 (0.03) | 0.62 (0.23) | 0.52 (0.09)

6. Secondary Outcome: Terminal Phase Half-life (t1/2) Everolimus
Description: Venous blood draw up to 24 hours prior to implantation of the first study stent (predose time point), at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours after completion of implantation of the last study stent.
Time Frame: Predose <24 hours; post dose at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours
Population: Analysis groups have ≥3 subjects. Everolimus concentrations declined rapidly in all subjects; half-life could be inaccurately determined for a subset of samples; determined by extrapolation of terminal phase. Concentrations not above detection limit in the terminal phase for enough time points for most subjects to accurately determine half-life.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Everolimus Dose of 95.4 µg | Everolimus Dose of 102.4 µg | Everolimus Dose of 138.6 µg
Number analyzed (Participants) | 4 | 7 | 3
Hours | 34.19 (20.81) | 22.83 (7.20) | 136.06 (62.08)

7. Secondary Outcome: Total Blood Clearance - Everolimus (CL)
Description: Venous blood draw up to 24 hours prior to implantation of the first study stent (predose time point), 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours after completion of implantation of the last study stent.
Time Frame: Predose <24 hours; post dose at 30 minutes, 1, 2, 4, 6, 12, 24, 48, and 72 hours
Population: Analysis groups have ≥3 subjects. Everolimus concentrations declined rapidly in all subjects; CL could be inaccurately determined for a subset of samples; determined by extrapolation of terminal phase. Concentrations not above detection limit in the terminal phase for enough time points for most subjects to accurately determine CL value.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Everolimus Dose of 95.4 µg | Everolimus Dose of 102.4 µg | Everolimus Dose of 138.6 µg
Number analyzed (Participants) | 4 | 7 | 3
L/h | 6445 (3924) | 8044 (1276) | 2511 (1073)

8. Secondary Outcome: All Death
Description: Number of participants no longer alive
Time Frame: 6 months
Population: Analysis was intention to treat; all patients in the study underwent clinical follow up to provide the information needed for this endpoint.
Measure: Number; unit: percentage of participants who died
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
percentage of participants who died | 0.0

9. Secondary Outcome: Myocardial Infarction (MI) Related to the Target Vessel
Description: New Q-waves in ≥2 leads lasting ≥0.04 sec with creatine kinase (CK) MB or troponin >normal; if no new Q-waves total CK levels >3× normal (peri-percutaneous coronary intervention [PCI]) or >2× normal (spontaneous) with elevated CK-MB or troponin >3× normal (peri-PCI) or >2× normal (spontaneous) plus at least one of the following: ECG changes indicating new ischemia (new ST-T changes, left bundle branch block), imaging evidence of new loss of viable myocardium, or new regional wall motion abnormality. Similar for MI diagnosis post coronary artery bypass graft with CK-MB or troponin >5× normal
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
percentage of participants | 0.0

10. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: TVR is any ischemia-driven repeat percutaneous intervention to improve blood flow, or bypass surgery of not previously existing lesions with diameter stenosis ≥50% by quantitative coronary angiography in the target vessel, including the target lesion.
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
percentage of participants | 0.0

11. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: TLR is any ischemia-driven repeat percutaneous intervention to improve blood flow of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion.
Time Frame: 6 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
percentage of participants | 0.0

12. Secondary Outcome: Definite + Probable Stent Thrombosis (ST) Rate Based on Academic Research Consortium (ARC) Definition
Description: DEFINITE ST: acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE ST: unexplained death within 30 days or target-vessel infarction without angiographic information ARC ST is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute ST: 0-24 hours after stent implantation; Subacute ST: >24 hours to 30 days post; late ST: >30 days to 1 year post; Very late ST: >1 year post; NOTE: Acute/subacute can be replaced by early ST (0-30 days).
Time Frame: 24 hours
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
percentage of participants | 0.0

13. Secondary Outcome: Definite + Probable Stent Thrombosis Rate Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 12
Time Frame: >24 hours-30 days
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
percentage of participants | 0.0

14. Secondary Outcome: Definite + Probable Stent Thrombosis Rate Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 12
Time Frame: >30 days-1 year
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 22
percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PROMUS Element
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=22)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=22)
Catheter site haematoma (General disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to Sponsor for review at least 45 days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.